CLINICAL TRIAL: NCT01490060
Title: Evaluation of Fosaprepitant's Effect on Drug Metabolism in Sarcoma Patients Receiving Ifosfamide-based Multi-day Chemotherapy Regimen
Brief Title: Fosaprepitant in Patients Receiving Ifosfamide-based Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0620; NCI-2012-00011 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Sarcoma; Chemotherapy-induced Nausea and Vomiting; Effects of Chemotherapy; Adverse Effects of Medical Drugs
Keywords: cancer; fosaprepitant; Ifosfamide-based Multi-day Chemotherapy; Chemotherapy-induced nausea and vomiting; CINV; multi-day chemotherapy regimens; antiemetics; adverse effect; doxorubicin plus ifosfamide; AI; AI and vincristine; VAI; aprepitant; prevention; nausea; vomiting; emetogenic chemotherapy
MeSH Terms: conditions — Sarcoma; Vomiting; Neoplasms; Nausea | interventions — fosaprepitant; Dexamethasone; dexamethasone acetate; Calcium Dobesilate; Doxorubicin; Mesna; Ifosfamide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Dose Day 1 (Experimental): Arm 1, Single Dose: Fosaprepitant 150 mg intravenous (IV) Day 1 of Cycle 1 or Day 1 of Cycle 2. Participants randomized to Group 1 (Fosaprepitant Cycle 1 + No Fosaprepitant Cycle 2); or Group 2 (No Fosaprepitant Cycle 1 and Fosaprepitant Cycle 2). Dexamethasone intravenously (IVPB) daily for 5 days (12 mg on day 1, and 8 mg on days 2-5) and 5HT3 receptor antagonist as standard of care 30 minutes prior to chemotherapy. Doxorubicin 25 mg/m^2/day IV continuous infusion for 72 hours on days 1, 2, and 3, completing infusion on day 4 (total dose: 75 mg/m^2) as part of AI Chemotherapy.
  Interventions: Drug: Fosaprepitant; Drug: Dexamethasone; Drug: 5HT3 receptor antagonist; Drug: Ifosfamide-based chemotherapy (AI); Drug: Doxorubicin; Drug: Mesna; Drug: Ifosfamide; Drug: Vincristine
- Two Doses Day 1 + Day 4 (Experimental): Arm 2, Two Doses: Fosaprepitant 150 mg IV Day 1 + Day 4 of Cycle 1 or Day 1 + Day 4 of Cycle 2. Participants randomized to Group 1 (Fosaprepitant Cycle 1 + No Fosaprepitant Cycle 2); or Group 2 (No Fosaprepitant Cycle 1 and Fosaprepitant Cycle 2). Dexamethasone intravenously (IVPB) daily for 5 days (12 mg on day 1, and 8 mg on days 2-5) and 5HT3 receptor antagonist as standard of care 30 minutes prior to chemotherapy. Doxorubicin 25 mg/m^2/day IV continuous infusion for 72 hours on days 1, 2, and 3, completing infusion on day 4 (total dose: 75 mg/m^2) as part of AI Chemotherapy.
  Interventions: Drug: Fosaprepitant; Drug: Dexamethasone; Drug: 5HT3 receptor antagonist; Drug: Ifosfamide-based chemotherapy (AI); Drug: Doxorubicin; Drug: Mesna; Drug: Ifosfamide; Drug: Vincristine

INTERVENTIONS:
Drug: Fosaprepitant — 150 mg administered intravenously, delivered in either single dose or two doses, on Day 1 for single dose and on Days 1 and 4 for two doses, varying between Cycle 1 or Cycle 2 depending upon randomization to arm.
  Other Names: Fosaprepitant Dimeglumine
Drug: Dexamethasone — Intravenous push (IVPB) daily for 5 days (12 mg on day 1, and 8 mg on days 2-5)
  Other Names: Dexamethasone acetate; Decadron
Drug: 5HT3 receptor antagonist — 5HT3 receptor antagonist as standard of care 30 minutes prior to chemotherapy
Drug: Ifosfamide-based chemotherapy (AI) — Doxorubicin + Mesna + + Ifosfamide + Vincristine, chemotherapy cycles repeated every 3-4 weeks for up to 6 cycles. Chemotherapy drugs listed separately, individual dosages, etc.
Drug: Doxorubicin — 25 mg/m^2/day IV continuous infusion for 72 hours on days 1, 2, and 3, completing infusion on day 4 (total dose: 75 mg/m^2) as part of AI Chemotherapy.
  Other Names: Rubex; Adriamycin; Adriamycin RDF; Adriamycin PFS; Doxorubicin Hydrochloride
Drug: Mesna — Prior to ifosfamide (Day 1) - 500 mg/m^2 (20% of ifosfamide dose) given simultaneously with ifosfamide and then daily continuous infusion (Days 1-4 completing infusion on day 4) - 1,500 mg/m^2/day (60% of daily ifosfamide dose) for a total of 6 gm/m^2. The mesna infusion complete 24 hours after last dose of ifosfamide.
  Other Names: Mesnex
Drug: Ifosfamide — 2.5 g/m^2 IV bolus over 3 hours on days 1, 2, 3, 4 (total dose: 10 g/m^2).
  Other Names: Ifex
Drug: Vincristine — 2 mg IV by rapid infusion (Day 1) may be given to participants with sarcomas of small cell histology.

SUMMARY:
The goal of this clinical research study is to learn how different doses of fosaprepitant may effect how ifosfamide-based chemotherapy is absorbed by the body. Researchers also want to learn if fosaprepitant can help to control or prevent delayed nausea and/or vomiting that may be caused by chemotherapy. The safety of this drug will also be studied.

Fosaprepitant is designed to block the natural substance in the brain that causes nausea and vomiting. This may help to prevent and/or control nausea and vomiting caused by chemotherapy.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will receive fosaprepitant during 21-day chemotherapy cycles. You will be randomly assigned (as in a toss of dice) to 1 of 2 study groups, each with 2 divisions:

* If you are in Group A1, you will receive fosaprepitant on Day 1 of Cycle 1.
* If you are in Group A2, you will receive fosaprepitant on Day 1 of Cycle 2.
* If you are in Group B1, you will receive fosaprepitant on Days 1 and 4 of Cycle 1.
* If you are in Group B2, you will receive fosaprepitant on Days 1 and 4 Cycle 2.

You and the study staff will know to which group and division you are assigned. Each time you receive the drug, you will receive it by vein over about 20-30 minutes.

You will also receive the ifosfamide-based chemotherapy prescribed by your doctor, as well as standard drugs for preventing nausea and vomiting (such as ondansetron, lorazepam, diphenhydramine, and promethazine). You will sign a separate consent form that will describe these treatments in detail, along with their risks.

You will receive dexamethasone before chemotherapy, every day for 5 days, to help prevent nausea and vomiting.

Before each chemotherapy cycle, you will be given a study diary. Each day, you will record any side effects you may . You should bring your study diary to every study visit so the study staff can review it.

Study Visits:

Before each cycle that you receive fosaprepitant, the following tests and procedures will be performed:

* You will have a physical exam.
* Your vital signs, weight, and performance status will be recorded.
* You will fill out the same questionnaire you did at screening.
* You will be asked about any other drugs you may be taking. Be sure to tell the study doctor about all drugs (including vitamins, herbal products, and nutritional supplements), because some drugs/substances will cause side effects when taken at the same time as fosaprepitant.
* Blood (about 5 teaspoons) will be drawn for routine tests.

Blood (about 1 teaspoon) will also be drawn 2 times each week during Cycles 1 and 2 for routine tests.

Pharmacokinetic Testing:

On Days 1 and 4 of Cycles 1 and 2 of chemotherapy, blood samples (about 2 teaspoons each time) will be drawn for pharmacokinetic (PK) testing, when possible. PK testing measures the amount of study drug in the body at different time points. The blood will be drawn before you receive ifosfamide, at the end of the infusion, and 4 more times in the 24 hours after the infusion.

Length of Study:

You may receive up to 6 cycles of chemotherapy (and up to 5 cycles of fosaprepitant). You will no longer be able to take the study drug if the disease gets worse or if intolerable side effects occur.

Your participation on the study will be over once you have completed the end-of-study visit.

End-of-Study Visit:

About 3 weeks after your last dose of fosaprepitant, you will return for an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam.
* Your vital signs, weight, and performance status will be recorded.
* You will fill out the same questionnaire you did at screening.
* You will be asked about any other drugs you may be taking.
* Blood (about 5 teaspoons) will be drawn for routine tests.

This is an investigational study. Fosaprepitant is FDA approved and commercially available in combination with other drugs for the prevention of nausea and vomiting that may be caused by chemotherapy. It is investigational to study how fosaprepitant may affect the drug levels of ifosfamide in the blood and how many doses should be given.

Up to 36 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sarcoma which is locally advanced, at high risk for relapse or metastatic for whom treatment with doxorubicin plus ifosfamide (AI) or AI and vincristine (VAI) is indicated.
2. Must be 18-65 years of age.
3. Male and Females of child bearing potential must use acceptable methods of birth control which include oral contraceptives, spermicide with either a condom, diaphragm or cervical cap, us of a intrauterine device (IUD) or abstinence.
4. Adequate hematologic (ANC >/= 1500/mm^3, platelet count >/= 100,000/mm^3), renal (serum creatinine </= 1.5 mg/dL), hepatic (serum bilirubin count </= 1.5 x normal and SGOT or SGPT </= 3 x normal) functions.
5. Karnofsky Performance Status >/= 60%
6. Signed informed consent form.
7. Patients are required to read and understand English to comply with protocol requirements.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with any co-morbid condition which renders patients at high risk of treatment complication.
3. Known allergy to fosaprepitant or any of its active components.
4. Patient has uncontrolled angina, congestive heart failure (New York Heart Association > class II or known ejection fraction < 40%), uncontrolled cardiac arrhythmia or hypertension, or acute myocardial infarction within 3 months.
5. Patient has an active seizure disorder. (Patients with a previous history of seizure disorders will be eligible for the study, if they have had no evidence of seizure activity, and they have been free of antiseizure medication for the previous 5 years).
6. Prior surgery or radiotherapy (RT) within 2 weeks of study entry.
7. Psychological, social, familial, or geographical reasons that would prevent scheduled visits and follow-up.
8. Patients receiving any medication for pre-existing nausea/vomiting will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 21, 2012 to January 23, 2014. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Arm A: Single Dose, Group 1: Fosaprepitant 150 mg intravenous (IV) Day 1 of Cycle 1 (Group 1). Participants Randomized to Group 1 (Fosaprepitant Cycle 1 + No Fosaprepitant Cycle 2). Dexamethasone IVPB daily for 5 days (12 mg on day 1, and 8 mg on days 2-5) and 5HT3 receptor antagonist as standard of care 30 min prior to chemotherapy. Doxorubicin 25 mg/m^2/day IV continuous infusion for 72 hrs on days 1, 2, and 3, completing infusion on day 4 (total dose: 75 mg/m^2). Mesna: Prior to ifosfamide (Day 1) - 500 mg/m^2 given simultaneously with ifosfamide and then daily CI (Days 1-4 completing infusion on day 4) - 1,500 mg/m^2/day for a total of 6 gm/m^2. The mesna infusion will complete 24 hrs after the last dose of ifosfamide. Ifosfamide: 2.5 g/m^2 IV bolus over 3 hrs on days 1, 2, 3, 4 (total dose: 10 g/m^2). Vincristine: 2 mg IV by rapid infusion (Day 1) may be given to participants with sarcomas of small cell histology.
- Arm A: Single Dose, Group 2: Fosaprepitant 150 mg intravenous (IV) Day 1 of Cycle 2 (Group 2). Participants Randomized to Group 2 (No Fosaprepitant Cycle 1 + Fosaprepitant Cycle 2). Dexamethasone IVPB daily for 5 days (12 mg on day 1, and 8 mg on days 2-5) and 5HT3 receptor antagonist as standard of care 30 min prior to chemotherapy. Doxorubicin 25 mg/m^2/day IV continuous infusion for 72 hrs on days 1, 2, and 3, completing infusion on day 4 (total dose: 75 mg/m^2). Mesna: Prior to ifosfamide (Day 1) - 500 mg/m^2 given simultaneously with ifosfamide and then daily CI (Days 1-4 completing infusion on day 4) - 1,500 mg/m^2/day for a total of 6 gm/m^2. The mesna infusion will complete 24 hrs after the last dose of ifosfamide. Ifosfamide: 2.5 g/m^2 IV bolus over 3 hrs on days 1, 2, 3, 4 (total dose: 10 g/m^2). Vincristine: 2 mg IV by rapid infusion (Day 1) may be given to participants with sarcomas of small cell histology.
- Arm B: Two Doses, Group 1: Fosaprepitant 150 mg IV Day 1 + Day 4 of Cycle 1 (Group 1). Participants Randomized to Group 1 (Fosaprepitant Cycle 1 + No Fosaprepitant Cycle 2). Dexamethasone IVPB daily for 5 days (12 mg on day 1, and 8 mg on days 2-5) and 5HT3 receptor antagonist as standard of care 30 min prior to chemotherapy. Doxorubicin 25 mg/m^2/day IV continuous infusion for 72 hrs on days 1, 2, and 3, completing infusion on day 4 (total dose: 75 mg/m^2). Mesna: Prior to ifosfamide (Day 1) - 500 mg/m^2 given simultaneously with ifosfamide and then daily CI (Days 1-4 completing infusion on day 4) - 1,500 mg/m^2/day for a total of 6 gm/m^2. The mesna infusion will complete 24 hrs after the last dose of ifosfamide. Ifosfamide: 2.5 g/m^2 IV bolus over 3 hrs on days 1, 2, 3, 4 (total dose: 10 g/m^2). Vincristine: 2 mg IV by rapid infusion (Day 1) may be given to participants with sarcomas of small cell histology.
- Arm B: Two Doses, Group 2: Fosaprepitant 150 mg IV Day 1 + Day 4 of Cycle 2 (Group 2). Participants Randomized to Group 2 (No Fosaprepitant Cycle 1 + Fosaprepitant Cycle 2). Dexamethasone IVPB daily for 5 days (12 mg on day 1, and 8 mg on days 2-5) and 5HT3 receptor antagonist as standard of care 30 min prior to chemotherapy. Doxorubicin 25 mg/m^2/day IV continuous infusion for 72 hrs on days 1, 2, and 3, completing infusion on day 4 (total dose: 75 mg/m^2). Mesna: Prior to ifosfamide (Day 1) - 500 mg/m^2 given simultaneously with ifosfamide and then daily CI (Days 1-4 completing infusion on day 4) - 1,500 mg/m^2/day for a total of 6 gm/m^2. The mesna infusion will complete 24 hrs after the last dose of ifosfamide. Ifosfamide: 2.5 g/m^2 IV bolus over 3 hrs on days 1, 2, 3, 4 (total dose: 10 g/m^2). Vincristine: 2 mg IV by rapid infusion (Day 1) may be given to participants with sarcomas of small cell histology.
Period: Cycle 1
Arm/Group | Arm A: Single Dose, Group 1 | Arm A: Single Dose, Group 2 | Arm B: Two Doses, Group 1 | Arm B: Two Doses, Group 2
Started | 11 | 13 | 12 | 11
Completed | 11 | 12 | 9 | 8
Not Completed | 0 | 1 | 3 | 3
Not completed — Change of Treatment | 0 | 1 | 1 | 1
Not completed — Insurance Denied | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Treatment at Another Facility | 0 | 0 | 0 | 1
Period: Cycle 2
Arm/Group | Arm A: Single Dose, Group 1 | Arm A: Single Dose, Group 2 | Arm B: Two Doses, Group 1 | Arm B: Two Doses, Group 2
Started | 11 | 12 | 9 | 8
Completed | 9 | 11 | 8 | 8
Not Completed | 2 | 1 | 1 | 0
Not completed — Change of Treatment | 1 | 1 | 0 | 0
Not completed — Non-Compliance | 0 | 0 | 1 | 0
Not completed — Adverse Event Related to Chemotherapy | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Single Dose, Day 1: Fosaprepitant 150 mg intravenous (IV) Day 1 of Cycle 1 (Group 1) or Day 1 of Cycle 2 (Group 2). Participants Randomized to Group 1 (Fosaprepitant Cycle 1 + No Fosaprepitant Cycle 2) or Group 2 (No Fosaprepitant Cycle 1 + Fosaprepitant Cycle 2).
- Arm B: Two Doses, Day 1 + Day 4: Fosaprepitant 150 mg IV Day 1 + Day 4 of Cycle 1 (Group 1) or Day 1 + Day 4 of Cycle 2 (Group 2). Participants Randomized to Group 1 (Fosaprepitant Cycle 1 + No Fosaprepitant Cycle 2) or Group 2 (No Fosaprepitant Cycle 1 + Fosaprepitant Cycle 2).
- Total: Total of all reporting groups
Arm/Group | Arm A: Single Dose, Day 1 | Arm B: Two Doses, Day 1 + Day 4 | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Customized [Number; unit: participants]
  Between 19 and 65 years | 24 | 23 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 16 | 13 | 29
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: Complete response (CR) defined as: No emetic episodes and no rescue medications. This is a cross-over designed study, the outcomes by single dose, two doses and control cycles were evaluated by combining the results from both cycle 1 and cycle 2 according to the treatment received.
Time Frame: From Day 1 to Day 5 in two 21-days cycles (Cycle 1 and Cycle 2).
Population: Out of 40 eligible participants, 2 participants had change of treatment, 1 participant was noncompliant and 1 participant had an adverse event related to chemotherapy. 36 participants completed cycle 1 and cycle 2.
Measure: Number; unit: percentage of participants
Groups:
- Control Cycle (Arm A/Arm B): Control cycle without fosaprepitant.
Arm/Group | Control Cycle (Arm A/Arm B) | Arm A: Single Dose, Day 1 | Arm B: Two Doses, Day 1 + Day 4
Number analyzed (Participants) | 36 | 20 | 16
percentage of participants | 17 | 10 | 50

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious Adverse Events (SAEs) were assessed in two 21-days cycles (Cycle 1 and Cycle 2). Collection period: May 23, 2012 to June 11, 2014.
Description: Number of participants for different study groups are: 22 single dose, Arm A (11 from group 1, cycle 1 & 11 from group 2, cycle 2); 17 two doses, Arm B (9 from group 1, cycle 1 & 8 from group 2, cycle 2); 37 control cycle [Arm A: 21(12 from group 1, cycle 2 & 11 from group 2,cycle 1); Arm B: 16(8 from group 1, cycle 2 & 8 from group 2,cycle 1)].
Arm/Group | Control Cycle (Arm A/Arm B) | Arm A: Single Dose, Day 1 | Arm B: Two Doses, Day 1 + Day 4
Serious Adverse Events (participants affected / at risk) | 4/37 | 1/22 | 1/17
Other Adverse Events (participants affected / at risk) | 35/37 | 22/22 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Cycle (Arm A/Arm B) (N=37) | Arm A: Single Dose, Day 1 (N=22) | Arm B: Two Doses, Day 1 + Day 4 (N=17)
Neutropenic Fever (General disorders) | 4 (4) | 1 (1) | 1 (1) — Related to Myelosuppression from chemotherapy in the first 2 cycles.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Cycle (Arm A/Arm B) (N=37) | Arm A: Single Dose, Day 1 (N=22) | Arm B: Two Doses, Day 1 + Day 4 (N=17)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 19 (19) | 9 (9) | 9 (9)
Anorexia (Gastrointestinal disorders) | 22 (22) | 12 (12) | 3 (3)
Fatigue (General disorders) | 25 (25) | 12 (12) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (4)
Chills (General disorders) | 7 (7) | 6 (6) | 5 (5)
Headache (General disorders) | 9 (9) | 5 (5) | 4 (4)
Memory Impairment (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2)
Paresthesia (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 2 (2)
Pain (General disorders) | 5 (5) | 4 (4) | 3 (3)
Alopecia (General disorders) | 10 (10) | 5 (5) | 1 (1)
Eye Disorders (Eye disorders) | 6 (6) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes